# Assessing the Impact of myHealth Rewards Enrollment Emails (NCT04047342)

## Study Protocol with Statistical Analysis Plan

December 7, 2020

### **Study Protocol**

## **Purpose**

The purpose of the study was to evaluate, prospectively, the potential impact of different email message conditions (standard promotional email and loss frame) on enrollment in a wellness program (myHealth Rewards) by Geisinger Health Plan (GHP) members who have recently been hired at Geisinger. The current study was developed to test whether the loss frame email was more effective than a standard reminder email, particularly for a population that was new to the organization. It was hypothesized that the loss frame email would increase enrollment more compared to the standard email.

#### Methods

## Sample

There were 831 new employees who received emails from July 16, 2019 to October 8, 2019. Enrollment data was gathered until December 20, 2019. Of these employees, 7 were excluded for registering before the emails were sent (e.g., after learning about the program during new hire orientation). The final sample consisted of 824 employees.

## **Control and experimental conditions**

**Standard Email.** The standard email mentioned the average premium savings, the speed and ease of starting the enrollment process, and the deadline for registering and having health measures on file. The standard email also provided two button links for registering and finding free health screenings where health measures could be collected and registered at one convenient time and location. This group served as the active control group.

Loss frame email. The loss frame email had a subject line suggesting that employees were currently "throwing away" a precise dollar amount by not participating and that they could therefore avoid missing out on substantial gains (i.e., savings) by taking action. This email contained and built upon all of the same information included in the standard email.

#### Outcome measures

The outcome measure was enrollment in the myHealth Rewards program. This measure was binary, and data was collected until December 20, 2019. Although the number of people who clicked on the link was planned as another primary outcome measure, this data was not collected due to administrative error.

## **Statistical Analysis Plan**

Binary logistic generalized linear models (GLMs) were used to analyze enrollment and as a function of experimental condition, with the standard email group as a reference group. Odds ratios (ORs) were calculated, along with 95% confidence intervals (CIs); two-tailed p-values < 0.05 were used to determine statistical significance. To represent effect size, the standardized statistic, Cohen's d, was estimated using the formula  $LogOddsRatio \times \sqrt{3}/\pi$  (Hasselblad & Hedges, 1995). Raw percentages with 95% CIs were also presented in graphs. All analyses were conducted in R.